CLINICAL TRIAL: NCT00003788
Title: Prospective Clinical Trials in the Use of Photodynamic Therapy (PDT) for the Treatment of Malignant Supratentorial Brain Tumors
Brief Title: Surgery, Radiation Therapy, and Chemotherapy With or Without Photodynamic Therapy in Treating Patients With Newly Diagnosed or Recurrent Malignant Supratentorial Gliomas
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Colorado Health Foundation (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066927; HEALTHONE-43892; HEALTHONE-1A; HEALTHONE-CA43892; RPCI-DS-9802; NCI-V99-1525
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2003-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — Carmustine; Lomustine; Dihematoporphyrin Ether; Procarbazine; Neoadjuvant Therapy; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Drug: carmustine
Drug: lomustine
Drug: porfimer sodium
Drug: procarbazine hydrochloride
Procedure: neoadjuvant therapy
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. It is not yet known if the addition of photodynamic therapy to combined therapy with surgery, radiation therapy, and chemotherapy is more effective than combined therapy alone for supratentorial gliomas.

PURPOSE: Randomized phase III trial to study the effectiveness of surgery, radiation therapy, and chemotherapy with or without photodynamic therapy in treating patients who have newly diagnosed or recurrent malignant supratentorial gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the addition of photodynamic therapy to standard brain tumor care (surgical resection, postoperative radiotherapy, and chemotherapy) will result in a significant prolongation of time to recurrence and survival in newly diagnosed malignant supratentorial gliomas.
* Compare the effect of high or low light dose photodynamic therapy on survival of patients with recurrent malignant supratentorial gliomas.

OUTLINE: This is a randomized, multicenter, two part study. Patients are stratified according to clinical center.

Newly diagnosed patients (Study 1)

* Patients are randomized to receive either high light dose photodynamic therapy (arm I) or no photodynamic therapy (arm II):

  * Arm I: Patients receive porfimer sodium (Photofrin) IV one day prior to surgery. Craniotomy and tumor resection are performed. Upon completion of resection, patients undergo intracavitary photoillumination with a high light dose.
  * Arm II: Craniotomy and tumor resection are performed. Postoperatively, all patients receive external beam radiotherapy 5 days per week for 5-6 weeks. After completing radiotherapy, patients receive nitrosourea (carmustine or lomustine) chemotherapy.

Recurrent tumor patients (Study 2)

* Patients receive Photofrin IV one day prior to surgery. Craniotomy and tumor resection are performed.

  * Arm I: Patients receive high dose light therapy during surgery.
  * Arm II: Patients receive low dose light therapy during surgery. Patients receive chemotherapy with procarbazine for 28 days beginning 2-4 weeks after surgery. Courses repeat every 56 days in the absence of disease progression or unacceptable toxicity.

Patients are followed on both studies at 4 weeks postsurgery, then every 3 months until death or for 1 year after study closure.

PROJECTED ACCRUAL: A minimum of 150 patients with newly diagnosed tumor will be accrued for this study within 4 years (Study 1). A maximum of 120 patients with recurrent disease will be accrued within 4.5 years (Study 2)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed or recurrent supratentorial glioblastoma or malignant astrocytoma

  * Grade 3 or 4 astrocytoma as defined by the Daumas-Duport classification
* Suitable for radical resection on the basis of imaging studies
* Patients with recurrent disease must have failed surgery and radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100% for newly diagnosed tumor
* Karnofsky 70-100% for recurrent tumor

Life expectancy:

* At least 3 months

Hematopoietic:

* Recurrent tumor:

  * WBC at least 2,000/mm^3
  * Platelet count at least 80,000/mm^3

Hepatic:

* Recurrent tumor:

  * PT/PTT no greater than 1.5 times upper limit of normal (ULN)
  * Bilirubin and LFTs less than 2 times ULN
  * Alkaline phosphatase no greater than 3 times ULN
  * GGT no greater than 3 times ULN

Renal:

* Creatinine no greater than 2 mg/dL

Other:

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior cranial radiotherapy for newly diagnosed tumor

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 1998-04

CONTACTS AND LOCATIONS:
Overall Officials: Fred W. Hetzel, PhD, JD, Study Chair — Colorado Health Foundation
Locations (4):
- United States (3):
  - Rocky Mountain Neurological Associates, Englewood, Colorado
  - Roswell Park Cancer Institute, Buffalo, New York
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
- St. Michael's Hospital-Annex, Toronto, Ontario, Canada